CLINICAL TRIAL: NCT03421054
Title: Pilot, Open Non-controled Trial to Assess the Feasibility of Implementing Objective Parameters as Primary Endpoints in a Clinical Trial With Patients Affected by Knee Osteoarthritis
Brief Title: Pilot Trial to Assess the Feasibility of Implementing Objective Parameters in Patients Affected by Knee Osteoarthritis
Acronym: SMILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: River Pharma S.r.l. (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pilot OPRPH/0117/FS
Record Dates: First submitted 2018-01-29; First posted 2018-02-05 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nutraceutical containing HA (Other): pain reduction of the affected knee in the patients assuming nutraceutical containing HA
  Interventions: Dietary Supplement: patients assuming nutraceutical containing HA

INTERVENTIONS:
Dietary Supplement: patients assuming nutraceutical containing HA — pain reduction of the affected knee in the patients assuming nutraceutical containing HA

SUMMARY:
Pilot, open non-controlled trial to assess the feasibility of implementing objective parameters as primary endpoints in a clinical trial with patients affected by knee osteoarthritis.

DETAILED DESCRIPTION:
• to assess the feasibility of implementing ultrasonography and Range of motion (ROM) as objective measurements to correlate the improvement of the knee mobility with the pain reduction of the affected knee in the patients assuming nutraceutical containing HA.

The secondary objectives of the trial are:

* to assess the feasibility of implementing Actigraphy as objective measurements to correlate the improvement of the knee mobility with the pain reduction (optional).
* to evaluate the enrollment range in one month.

The explorative objectives of the trial are:

• Preliminary data on efficacy of the tested product

ELIGIBILITY:
Inclusion Criteria:

* Any gender and age from 50 to 70 years
* Symptomatic osteoarthritis (OA) of the knee with mild joint discomfort for at least 6 months prior to enrollment, following ACR criteria with history and physical examination (1). Subjects diagnosed with bilateral knee OA will be asked to specify the most affected knee at baseline, and this knee will be evaluated throughout the study period.
* Available confirmatory X-ray (performed within the previous 6 months) diagnosis (Kellgren/Lawrence score 2) at the evaluated knee joint (2).
* Subjects experienced pain for at least 15 of the 30 days prior to the start of the study.

Exclusion Criteria:

* Subjects who have any inflammatory arthritic condition (different from the OA of the knee), fibromyalgia, multiple sclerosis or autoimmune disorder.
* Treatment with oral corticosteroids within 4 weeks before screening.
* Intra-articular injections of HA or corticosteroids in the target joint within 3 months before screening.
* Treatment with anti-inflammatory or chondroprotective drugs (chondroitin sulfate, glucosamine, methylsulfonylmethane, HA, diacerein) 2 weeks before the selection.
* HA-containing nutritional supplements or cosmetics during the month before the study.
* Previous surgical treatment of knee joint(s) or its necessity; complication(s) necessary for hospitalization and surgical treatment.
* Significant injury to the target joint within the past 6 months prior to screening (identified from medical history).
* Subjects following an energy-restricted diet for weight loss.
* Pregnant women, nursing mothers, or women (only if childbearing potential) not using adequate methods of contraception.
* Subjects with cardiovascular, hepatic, renal, respiratory, or hematologic illness, or other medical or psychiatric condition that, in the opinion of the investigator, would compromise participation or be likely to lead to hospitalization during the course of the study.
* Participation in an interventional clinical study in the previous 30 days.
* Presence of any clinically significant medical condition judged by the investigator to preclude the patient's inclusion in the study.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-04-15 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
synovial effusion reduction | week 4 and 8
  Correlation between reduction in VAS (at rest) and ultrasonography parameters

SECONDARY OUTCOMES:
pain reduction | week 4 and 8
  Correlation between reduction in VAS (at rest; on moving; on pressing) and Actigraphy parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan Andor, MD, Principal Investigator — MEDICALI'S
Locations (1):
- Opera Contract Research Organization S.r.l., Timișoara, Timiș County, Romania

REFERENCES:
- [Background] Bhatia D, Bejarano T, Novo M. Current interventions in the management of knee osteoarthritis. J Pharm Bioallied Sci. 2013 Jan;5(1):30-8. doi: 10.4103/0975-7406.106561. PMID 23559821
- [Background] Carvalho NA, Bittar ST, Pinto FR, Ferreira M, Sitta RR. Manual for guided home exercises for osteoarthritis of the knee. Clinics (Sao Paulo). 2010 Jun;65(8):775-80. doi: 10.1590/s1807-59322010000800006. PMID 20835554
- [Background] Voelker R. Few adults with knee osteoarthritis meet national guidelines for physical activity. JAMA. 2011 Oct 5;306(13):1428, 1430. doi: 10.1001/jama.2011.1388. No abstract available. PMID 21972300
- [Background] Pai YC, Chang HJ, Chang RW, Sinacore JM, Lewis JL. Alteration in multijoint dynamics in patients with bilateral knee osteoarthritis. Arthritis Rheum. 1994 Sep;37(9):1297-304. doi: 10.1002/art.1780370905. PMID 7945492
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Cutolo M, Berenbaum F, Hochberg M, Punzi L, Reginster JY. Commentary on recent therapeutic guidelines for osteoarthritis. Semin Arthritis Rheum. 2015 Jun;44(6):611-7. doi: 10.1016/j.semarthrit.2014.12.003. Epub 2014 Dec 24. PMID 25677861
- [Background] Bruyere O, Cooper C, Pelletier JP, Branco J, Luisa Brandi M, Guillemin F, Hochberg MC, Kanis JA, Kvien TK, Martel-Pelletier J, Rizzoli R, Silverman S, Reginster JY. An algorithm recommendation for the management of knee osteoarthritis in Europe and internationally: a report from a task force of the European Society for Clinical and Economic Aspects of Osteoporosis and Osteoarthritis (ESCEO). Semin Arthritis Rheum. 2014 Dec;44(3):253-63. doi: 10.1016/j.semarthrit.2014.05.014. Epub 2014 May 14. PMID 24953861
- [Background] Bruyere O, Burlet N, Delmas PD, Rizzoli R, Cooper C, Reginster JY. Evaluation of symptomatic slow-acting drugs in osteoarthritis using the GRADE system. BMC Musculoskelet Disord. 2008 Dec 16;9:165. doi: 10.1186/1471-2474-9-165. PMID 19087296
- [Background] Bannuru RR, Schmid CH, Kent DM, Vaysbrot EE, Wong JB, McAlindon TE. Comparative effectiveness of pharmacologic interventions for knee osteoarthritis: a systematic review and network meta-analysis. Ann Intern Med. 2015 Jan 6;162(1):46-54. doi: 10.7326/M14-1231. PMID 25560713
- [Background] Navarro-Sarabia F, Coronel P, Collantes E, Navarro FJ, de la Serna AR, Naranjo A, Gimeno M, Herrero-Beaumont G; AMELIA study group. A 40-month multicentre, randomised placebo-controlled study to assess the efficacy and carry-over effect of repeated intra-articular injections of hyaluronic acid in knee osteoarthritis: the AMELIA project. Ann Rheum Dis. 2011 Nov;70(11):1957-62. doi: 10.1136/ard.2011.152017. Epub 2011 Aug 17. PMID 21852252
- [Background] Waddell DD, Bricker DC. Total knee replacement delayed with Hylan G-F 20 use in patients with grade IV osteoarthritis. J Manag Care Pharm. 2007 Mar;13(2):113-121. doi: 10.18553/jmcp.2007.13.2.113. PMID 17330972
- [Background] Reed RK, Townsley MI, Laurent TC, Taylor AE. Hyaluronan flux from cat intestine: changes with lymph flow. Am J Physiol. 1992 Feb;262(2 Pt 2):H457-62. doi: 10.1152/ajpheart.1992.262.2.H457. PMID 1539704
- [Background] Balogh L, Polyak A, Mathe D, Kiraly R, Thuroczy J, Terez M, Janoki G, Ting Y, Bucci LR, Schauss AG. Absorption, uptake and tissue affinity of high-molecular-weight hyaluronan after oral administration in rats and dogs. J Agric Food Chem. 2008 Nov 26;56(22):10582-93. doi: 10.1021/jf8017029. PMID 18959406
- [Background] Hisada N, Satsu H, Mori A, Totsuka M, Kamei J, Nozawa T, Shimizu M. Low-molecular-weight hyaluronan permeates through human intestinal Caco-2 cell monolayers via the paracellular pathway. Biosci Biotechnol Biochem. 2008 Apr;72(4):1111-4. doi: 10.1271/bbb.70748. Epub 2008 Apr 7. PMID 18391466
- [Background] Laznicek M, Laznickova A, Cozikova D, Velebny V. Preclinical pharmacokinetics of radiolabelled hyaluronan. Pharmacol Rep. 2012;64(2):428-37. doi: 10.1016/s1734-1140(12)70784-3. PMID 22661195
- [Background] Altman RD, Manjoo A, Fierlinger A, Niazi F, Nicholls M. The mechanism of action for hyaluronic acid treatment in the osteoarthritic knee: a systematic review. BMC Musculoskelet Disord. 2015 Oct 26;16:321. doi: 10.1186/s12891-015-0775-z. PMID 26503103
- [Background] du Souich P. Absorption, distribution and mechanism of action of SYSADOAS. Pharmacol Ther. 2014 Jun;142(3):362-74. doi: 10.1016/j.pharmthera.2014.01.002. Epub 2014 Jan 21. PMID 24457028
- [Background] Oe M, Tashiro T, Yoshida H, Nishiyama H, Masuda Y, Maruyama K, Koikeda T, Maruya R, Fukui N. Oral hyaluronan relieves knee pain: a review. Nutr J. 2016 Jan 27;15:11. doi: 10.1186/s12937-016-0128-2. PMID 26818459
- [Background] Yasui T, Akatsuka M, Tobetto K, Hayaishi M, Ando T. The effect of hyaluronan on interleukin-1 alpha-induced prostaglandin E2 production in human osteoarthritic synovial cells. Agents Actions. 1992 Sep;37(1-2):155-6. doi: 10.1007/BF01987905. PMID 1456177
- [Background] Homandberg GA, Ummadi V, Kang H. The role of insulin-like growth factor-I in hyaluronan mediated repair of cultured cartilage explants. Inflamm Res. 2004 Aug;53(8):396-404. doi: 10.1007/s00011-004-1276-y. Epub 2004 Aug 10. PMID 15316671
- [Background] Wang CT, Lin YT, Chiang BL, Lin YH, Hou SM. High molecular weight hyaluronic acid down-regulates the gene expression of osteoarthritis-associated cytokines and enzymes in fibroblast-like synoviocytes from patients with early osteoarthritis. Osteoarthritis Cartilage. 2006 Dec;14(12):1237-47. doi: 10.1016/j.joca.2006.05.009. Epub 2006 Jun 30. PMID 16806998
- [Background] Waller KA, Zhang LX, Fleming BC, Jay GD. Preventing friction-induced chondrocyte apoptosis: comparison of human synovial fluid and hylan G-F 20. J Rheumatol. 2012 Jul;39(7):1473-80. doi: 10.3899/jrheum.111427. Epub 2012 Jun 1. PMID 22660808
- [Background] Bernad Pineda M. Current status of symptomatic slow-acting drugs for osteoarthritis (SYSADOAs) in Spain. Reumatol Clin. 2016 Jul-Aug;12(4):181-3. doi: 10.1016/j.reuma.2016.03.012. Epub 2016 Apr 18. No abstract available. English, Spanish. PMID 27101743
- [Background] Tashiro T, Seino S, Sato T, Matsuoka R, Masuda Y, Fukui N. Oral administration of polymer hyaluronic acid alleviates symptoms of knee osteoarthritis: a double-blind, placebo-controlled study over a 12-month period. ScientificWorldJournal. 2012;2012:167928. doi: 10.1100/2012/167928. Epub 2012 Nov 20. PMID 23226979
- [Background] Nagaoka I, Nabeshima K, Murakami S, Yamamoto T, Watanabe K, Tomonaga A, Yamaguchi H. Evaluation of the effects of a supplementary diet containing chicken comb extract on symptoms and cartilage metabolism in patients with knee osteoarthritis. Exp Ther Med. 2010 Sep;1(5):817-827. doi: 10.3892/etm.2010.114. Epub 2010 Jul 12. PMID 22993606
- [Background] D'Agostino MA, Conaghan P, Le Bars M, Baron G, Grassi W, Martin-Mola E, Wakefield R, Brasseur JL, So A, Backhaus M, Malaise M, Burmester G, Schmidely N, Ravaud P, Dougados M, Emery P. EULAR report on the use of ultrasonography in painful knee osteoarthritis. Part 1: prevalence of inflammation in osteoarthritis. Ann Rheum Dis. 2005 Dec;64(12):1703-9. doi: 10.1136/ard.2005.037994. Epub 2005 May 5. PMID 15878903
- [Background] Hartung W, Kellner H, Strunk J, Sattler H, Schmidt WA, Ehrenstein B, Fleck M, Backhaus M. Development and evaluation of a novel ultrasound score for large joints in rheumatoid arthritis: one year of experience in daily clinical practice. Arthritis Care Res (Hoboken). 2012 May;64(5):675-82. doi: 10.1002/acr.21574. PMID 22183834
- [Background] Serban O, Porojan M, Deac M, Cozma F, Solomon C, Lenghel M, Micu M, Fodor D. Pain in bilateral knee osteoarthritis - correlations between clinical examination, radiological, and ultrasonographical findings. Med Ultrason. 2016 Sep;18(3):318-25. doi: 10.11152/mu.2013.2066.183.pin. PMID 27622408
- [Background] Wu PT, Shao CJ, Wu KC, Wu TT, Chern TC, Kuo LC, Jou IM. Pain in patients with equal radiographic grades of osteoarthritis in both knees: the value of gray scale ultrasound. Osteoarthritis Cartilage. 2012 Dec;20(12):1507-13. doi: 10.1016/j.joca.2012.08.021. Epub 2012 Sep 1. PMID 22944523
- [Background] Yoshimura M, Aoba Y, Watari T, Momomura R, Watanabe K, Tomonaga A, Matsunaga M, Suda Y, Lee WY, Asai K, Yoshimura K, Nakagawa T, Yamamoto T, Yamaguchi H, Nagaoka I. Evaluation of the effect of a chicken comb extract-containing supplement on cartilage and bone metabolism in athletes. Exp Ther Med. 2012 Oct;4(4):577-580. doi: 10.3892/etm.2012.646. Epub 2012 Jul 24. PMID 23170108
- [Background] Yang CC, Hsu YL. A review of accelerometry-based wearable motion detectors for physical activity monitoring. Sensors (Basel). 2010;10(8):7772-88. doi: 10.3390/s100807772. Epub 2010 Aug 20. PMID 22163626
- [Background] Steins D, Dawes H, Esser P, Collett J. Wearable accelerometry-based technology capable of assessing functional activities in neurological populations in community settings: a systematic review. J Neuroeng Rehabil. 2014 Mar 13;11:36. doi: 10.1186/1743-0003-11-36. PMID 24625308
- [Background] Trudeau J, Van Inwegen R, Eaton T, Bhat G, Paillard F, Ng D, Tan K, Katz NP. Assessment of pain and activity using an electronic pain diary and actigraphy device in a randomized, placebo-controlled crossover trial of celecoxib in osteoarthritis of the knee. Pain Pract. 2015 Mar;15(3):247-55. doi: 10.1111/papr.12167. Epub 2014 Feb 5. PMID 24494935
- [Background] Wylde V, Lenguerrand E, Brunton L, Dieppe P, Gooberman-Hill R, Mann C, Blom AW. Does measuring the range of motion of the hip and knee add to the assessment of disability in people undergoing joint replacement? Orthop Traumatol Surg Res. 2014 Apr;100(2):183-6. doi: 10.1016/j.otsr.2013.09.016. Epub 2014 Feb 17. PMID 24556210
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Derived] Dogaru DE, Rosu S, Barattini DF, Guadagna S, Barattini L, Andor B. Assessment of the Feasibility of Objective Parameters as Primary End Points for Patients Affected by Knee Osteoarthritis: Protocol for a Pilot, Open Noncontrolled Trial (:SMILE:). JMIR Res Protoc. 2024 Jun 28;13:e13642. doi: 10.2196/13642. PMID 38941599
- See also: 46. Proverb resources: Ashanti Proverbs from Ghana — http://cogweb.ucla.edu/Discourse/Proverbs/Ashanti.html